CLINICAL TRIAL: NCT05733611
Title: A Phase 2 Clinical Trial Investigating Oncolytic Immunotherapy in Combination With Atezolizumab and Bevacizumab for the Treatment of Patients With Advanced Microsatellite Stable and Mismatch Repair Proficient Colorectal Carcinoma
Brief Title: RP2/RP3 in Combination With Atezolizumab and Bevacizumab for the Treatment of Patients With CRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons.
Sponsor: Replimune Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPL-004
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Refractory Metastatic Colorectal Cancer; pMMR; MSS
Keywords: Colorectal Carcinoma; Immunotherapy; Immuno-oncology; Oncolytic virus; Oncolytic immuno-gene therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RP2 and atezolizumab plus bevacizumab in advanced MSS and pMMR CRC (Experimental): RP2 will be injected by direct (including via colonoscope) or image-guided injection into injectable tumors (including subcutaneous, visceral, and nodal tumors).
  Interventions: Biological: RP2; Biological: atezolizumab; Biological: bevacizumab
- RP3 and atezolizumab plus bevacizumab in advanced MSS and pMMR CRC (Experimental): RP3 will be injected by direct (including via colonoscope) or image-guided injection into injectable tumors (including subcutaneous, visceral, and nodal tumors).
  Interventions: Biological: RP3; Biological: atezolizumab; Biological: bevacizumab

INTERVENTIONS:
Biological: RP2 — Genetically modified herpes simplex type 1 virus
  Arms: RP2 and atezolizumab plus bevacizumab in advanced MSS and pMMR CRC
Biological: RP3 — Genetically modified herpes simplex type 1 virus
  Arms: RP3 and atezolizumab plus bevacizumab in advanced MSS and pMMR CRC
Biological: atezolizumab — anti-PD-L1 monoclonal antibody
Biological: bevacizumab — anti-VEGF therapy

SUMMARY:
This is an open-label, Phase 2 clinical trial evaluating therapy with an oncolytic immunotherapy (RP2 or RP3) in combination with atezolizumab and bevacizumab in patients with advanced Microsatellite Stable and Mismatch Repair Proficient Colorectal Carcinoma.

DETAILED DESCRIPTION:
RP2 and RP3 are selectively replication competent herpes simplex viruses 1 (HSV-1) that express exogenous genes (RP2: GM-CSF, GALV, and anti-CTLA-4; RP3: GALV, and anti-CTLA-4 hCD40L, and h4-1BBL) intended for direct injection into suitable nonneurological solid tumors. They are genetically engineered to provide direct oncolytic tumor destruction combined with the induction of a systemic antitumor immune response.

This study will evaluate whether the use of oncolytic immunotherapy, either with RP2 or RP3, can provide meaningful efficacy in combination with an anti-PD-L1 therapy (atezolizumab) and anti-VEGF therapy (bevacizumab) in patients with advanced MSS and pMMR CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Histological or cytologic diagnosis of colorectal adenocarcinoma that is unresectable or metastatic.
3. Have had disease progression or were intolerant to treatment protocols that included irinotecan and oxaliplatin. Epidermal growth factor receptor (EGFR) or vascular endothelial growth factor receptor (VEGFR) directed therapies are allowed as part of the previous therapy if indicated.
4. Has at least 1 measurable tumor of ≥1 cm in longest diameter (or ≥1.5cm shortest diameter for lymph nodes).
5. Has injectable tumor(s) of at least 1cm in aggregate total diameter.
6. Must be willing to consent to provide archival tumor biopsy samples obtained within 90 days prior to Screening, or a fresh tumor biopsy collected on Day 1 of treatment or earlier.
7. Has adequate hematologic function, including:

   * White blood cell count ≥2.0 × 10^9/L
   * Absolute neutrophil count ≥1.5 × 10^9/L
   * Platelet count ≥75 × 10^9/L
   * Hemoglobin ≥8 g/dL(transfusions allowed; however, patient must not be transfusion-dependent).
8. Has adequate hepatic function, including:

   * Total bilirubin ≤1.5 × upper limit of normal (ULN; except patients with Gilbert syndrome or liver metastases, who must have a total bilirubin of <2.0 × ULN)
   * Serum albumin ≥2.8 g/dL
   * Aspartate aminotransferase and alanine aminotransferase (ALT)≤3.0 × ULN (or ≤5.0 × ULN, if liver metastases are present).
9. Has adequate renal function, defined as serum creatinine ≤1.5 × ULN or creatinine clearance ≥30 mL/minute (measured using Cockcroft-Gault formula or by 24-hour urine collection).
10. Prothrombin time ≤1.5 × ULN (or international normalization ratio [INR] ≤1.3) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN.

    Note: Patients who are on chronic anticoagulant therapy may be enrolled if the pretreatment INR<2.5. For patients requiring a deep injection of RP2/RP3, the INR must be <1.5 at the time of injection.
11. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1.
12. Female and male patients of reproductive potential must agree to avoid becoming pregnant or impregnating a partner and adhere to highly effective contraception requirements during the treatment period and for at least (a) 90 days after the last dose of RP2 or RP3 or (b) 5 months after the last dose of atezolizumab or (c) 6 months after the last dose of bevacizumab, whichever is longer.
13. Women of childbearing potential must have a negative serum beta-human chorionic human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units of β-hCG within 72 hours before the first dose and a negative urine pregnancy test on D-1.
14. Capable of giving signed informed consent which includes willingness to comply with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Prior treatment with regorafenib, trifluridine/tipiracil, fruquintinib, and immunotherapies.
2. Has received more than 3 lines of therapy for CRC.
3. Has microsatellite instability-high (MSI-H)/deficient DNA mismatch repair (dMMR)disease or BRAF V600E mutation.
4. Acute or chronic hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or acute or chronic hepatitis C virus (HCV; defined as HCV RNA [qualitative] is detected).

   Note: Patients who have been effectively treated are eligible for enrollment. Patients must be negative for HBsAg and HCV RNA.
5. Known human immunodeficiency virus (HIV) infection.

   Note: Testing for HIV is not required unless mandated by local health authority or clinically indicated.
6. Had systemic infection requiring intravenous (IV) antibiotics or other serious infection within 14 days prior to dosing.
7. With active significant herpetic infections or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis).

   Note: Patients with sporadic cold sores may be enrolled as long as no active cold sores are present at the time of Day 1
8. Active or history of central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Prior malignancy active within the previous 3 years, except for locally curable cancers that have apparently been cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
10. Macroscopic intravascular invasion into any large blood vessel such as the main portal vein, hepatic vein, pulmonary arteries or veins, aorta, or vena cava.
11. Had a significant bleeding event within the last 12 months that places the patient at unjustifiable risk for bleeding from deep intratumoral injection procedures based on Investigator assessment or interventional radiologist assessment.
12. History of significant cardiac vascular disease including myocarditis or congestive heart failure (defined as New York Heart Association Functional Classification III or IV), or unstable angina, serious uncontrolled cardiac arrhythmia, or myocardial infarction within 6 months of randomization.
13. Uncontrolled infection.
14. History or evidence of psychiatric disease, substance abuse, or any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the Investigator or the Medical Monitor, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.
15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
16. Active, known, or suspected autoimmune disease such as autoimmune thyroiditis and colitis requiring systemic immunomodulatory treatment. Note: Patients with diabetes mellitus, dysthyroidism without an autoimmune mechanism, and rheumatoid arthritis that do not require immunomodulatory treatment are permitted to enroll.
17. History of drug-induced interstitial lung disease, (noninfectious) pneumonitis that required steroids, or currently has pneumonitis.
18. Requires intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).
19. Has received a live vaccine within 28 days prior to the first dose of study treatment. Note: Seasonal influenza vaccines for injection or SARS-CoV-2 are generally inactivated vaccines and are allowed (See Section6.11.2for additional guidance). Live/attenuated vaccines (such as the intranasal influenza vaccines) are not allowed.
20. Is currently participating in or has participated in a study of an investigational agent within 4 weeks prior to the first dose of study treatment.

    Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks or 5 half-lives of the agent, whichever is longer, after the last dose of the previous investigational agent.
21. Conditions requiring treatment with immunosuppressive medications within 30 days. Inhaled or topical steroids, and adrenal replacement steroid dose are permitted in the absence of active autoimmune disease.

    Note: Patients who require a brief course (≤7 days) of corticosteroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. Physiologic replacement doses of systemic corticosteroids are permitted, only if the dose does not exceed 10 mg/day prednisone equivalent.
22. Conditions in which anticoagulant therapies cannot be safely stopped in the periprocedural period or patients on coumadin with a target INR >2.5 or that cannot be temporarily reversed to INR ≤1.7.
23. Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to treatment.
24. Prior organ transplantation including allogenic stem-cell transplantation.
25. Bowel obstruction, Major surgery ≤28 days prior to starting bevacizumab or anticipated major surgery while on study.

    Note: If a patient received major surgery, they must have recovered adequately prior to starting study treatment and must have adequate wound healing, based on Investigator's assessment or surgeon's assessment, before starting bevacizumab.
26. History of life-threatening toxicity related to prior immune therapy (eg, anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways [eg, CD40, 4-1BB]) except those that are unlikely to recur or are expected to be manageable with standard countermeasures (eg, hormone replacement after adrenal crisis). Individual cases should be discussed with a Medical Monitor if needed.
27. Presence of peritoneal disease, or lesions that are > 5 cm or liver tumors that are estimated to invade more than one-third of the liver.
28. Prior chemoembolization, radioembolization, or other locoregional liver-directed procedures to the lesion(s)selected for intratumoral injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From Day 1 to documented progression of disease (up to 3 years)
  Percentage of subjects achieving objective response (complete response + partial response).

SECONDARY OUTCOMES:
Frequency, Nature, and Severity of TEAEs and SAEs | From Screening through 60 days after last dose of RP2/RP3, or 135 days after last dose of atezolizumab/bevacizumab
  Percentage of subjects with TEAEs and SAEs
Overall Survival | From Day 1 to date of death by any cause (up to 3 years)
  Overall survival is defined as the time from the first day of study treatment to the date of death by any cause
Progression-free Survival | From Day 1 to documented progression of disease (up to 3 years)
  Progression-free survival is defined as the time from the first day of study treatment to the date of progression of disease, which was subsequently confirmed, or death by any cause, whichever occurs first
Duration of Response | From documented response to documented progression of disease (up to 3 years)
  Duration of response is defined as the time from documented response until the date of progression of disease, which was subsequently confirmed or with no further follow-up, or death due to any cause, whichever occurs first
Duration of Clinical Benefit | From Day 1 to loss of clinical benefit (up to 3 years)
  Duration of clinical benefit is defined as the time from the first day of study treatment to last progression of disease, which was subsequently confirmed or with no further follow-up for response, or death due to any cause, whichever occurs first, for subjects who achieve complete response, partial response, or stable disease
Complete Response Rate | From Day 1 to documented progression of disease (up to 3 years)
  Percentage of subjects achieving a complete response

CONTACTS AND LOCATIONS:
Overall Officials: Gary Vanasse, MD, Study Director — Replimune Inc.
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington